CLINICAL TRIAL: NCT02947100
Title: Phase I/II Safety and Dose Escalation Trial of the Omega-3 Fatty Acids Docosahexaenoic Acid (DHA) and Eicosapentaenoic Acid (EPA) in Children and Young Adults With Sickle Cell Disease (SCD)
Brief Title: Omega-3 Fatty Acids in Sickle Cell Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: manufacturing problem with study drug
Sponsor: Robin E. Miller (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); Thomas Jefferson University (Other); Solutex GC S.L. (Industry)
Responsible Party: Sponsor-Investigator, Robin E. Miller, Physician, Nemours Children's Clinic
Organization: Nemours Children's Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RM002; P20GM109021 (NIH)
Record Dates: First submitted 2016-10-18; First posted 2016-10-27 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; omega-3 fatty acids; Docosahexaenoic Acid (DHA); Eicosapentaenoic Acid (EPA)
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SCD-Omegatex™ (Experimental): single arm
  Interventions: Drug: SCD-Omegatex™

INTERVENTIONS:
Drug: SCD-Omegatex™ — Subjects will receive SCD-Omegatex™ (Enteric Fish Oil 250 DHA/27 EPA Soft Gelatin Capsule, 450 mg) at one of two daily doses, orally, once a day for 6 months. The trial will follow a "3+3" design using two dose levels. In the phase I portion, subjects will be treated with a dose of 25 mg/kg/day DHA and EPA. If this is tolerated without dose limiting toxicity (DLT), a subsequent cohort of patients will be treated at a dose of 37.5 mg/kg/day with a maximum total daily dose of 4 grams. Once a maximum tolerated dose (MTD) is determined, subjects on the phase II portion of the study will be treated at that dose.
  Other Names: Enteric Fish Oil 250 DHA/27 EPA Soft Gelatin Capsule

SUMMARY:
The purpose of this study is to determine the safety of a new formulation of the omega-3 fatty acids Docosahexaenoic Acid (DHA) and Eicosapentaenoic Acid (EPA) and to assess whether it decreases inflammation and inflammatory pain in children and young adults with Sickle Cell Disease.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria are eligible for enrollment into the study:

* Participant has signed the informed consent/assent with parent signing informed consent as age appropriate.
* Established diagnosis of HbSS, HbSC or HbSβo Thalassemia
* History of ≥1 vasoocclusive events (managed at home and/or in hospital) in preceding 12 months.
* Regular compliance with comprehensive care.
* Aged 8 years or greater and less than 26 years.
* At enrollment, subject should be in his/her baseline steady state and not in the midst of any acute complication due to SCD. Must be at least 2 weeks from infection or vasoocclusive crisis at time of screening labs

Exclusion Criteria:

* Baseline hemoglobin levels <5.5 gm/dL.
* Inability to swallow capsules
* Poor compliance with previous treatment regimens.
* Hepatic dysfunction
* Renal dysfunction
* PT and/or PTT ≥ 20% outside of normal
* Allergy to fish, shell fish or soy
* Triglyceride levels <80mg/dL.
* Pregnancy.
* Chronic Transfusion Therapy.
* Transfusion within the last 30 days.
* Treatment with any investigational drug or regular fish oil supplementations in last 60 days.
* Currently receiving another investigational agent, or on such an agent with the last 60 days.
* Dosage changes in preceding 3 months if on hydroxyurea
* Diagnosed bleeding disorder or patient on concomitant anti-coagulation.
* Conditional or abnormal result on most recent transcranial doppler or history of stroke.
* Other active chronic illness that could adversely affect subjects performance
* Children in Care
* Platelet count less than 100,000

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin E Miller, MD, Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours/Alfred I duPont Hospital for Children, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daak AA, Ghebremeskel K, Hassan Z, Attallah B, Azan HH, Elbashir MI, Crawford M. Effect of omega-3 (n-3) fatty acid supplementation in patients with sickle cell anemia: randomized, double-blind, placebo-controlled trial. Am J Clin Nutr. 2013 Jan;97(1):37-44. doi: 10.3945/ajcn.112.036319. Epub 2012 Nov 28. PMID 23193009
- [Background] Serhan CN. Resolution phase of inflammation: novel endogenous anti-inflammatory and proresolving lipid mediators and pathways. Annu Rev Immunol. 2007;25:101-37. doi: 10.1146/annurev.immunol.25.022106.141647. PMID 17090225
- [Background] Calder PC. Marine omega-3 fatty acids and inflammatory processes: Effects, mechanisms and clinical relevance. Biochim Biophys Acta. 2015 Apr;1851(4):469-84. doi: 10.1016/j.bbalip.2014.08.010. Epub 2014 Aug 20. PMID 25149823
- [Background] Tomer A, Kasey S, Connor WE, Clark S, Harker LA, Eckman JR. Reduction of pain episodes and prothrombotic activity in sickle cell disease by dietary n-3 fatty acids. Thromb Haemost. 2001 Jun;85(6):966-74. PMID 11434703

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SCD-Omegatex™
Started | 4
Completed | 0
Not Completed | 4
Not completed — study terminated early | 3
Not completed — did not meet inclusion criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | SCD-Omegatex™
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Clinical Safety, in a Dose Escalation Trial of SCD-Omegatex™ as Evidenced by an Absence of Adverse Events.
Description: No results are available from any outcome measures as study was stopped early due to manufacturing issues with study drug and will not be reopened.
Time Frame: 6 months with continuous monitoring
Population: Study was stopped early, before outcomes could be measured, due to manufacturing issues with the study drug
Arm/Group | SCD-Omegatex™
Number analyzed (Participants) | 0

2. Primary Outcome: Determine Whether 6 Months of Supplementation With SCD-Omegatex™ Will Reduce Thermal Sensitivity by Quantitative Sensory Testing to Below Pre-treatment Levels
Description: as for outcome 1
Time Frame: 6 months
Population: Study was stopped early, before outcomes could be measured, due to manufacturing issues with the study drug
Arm/Group | SCD-Omegatex™
Number analyzed (Participants) | 0

3. Secondary Outcome: Health-associated Quality of Life
Description: as for outcome 1
Time Frame: 6 months
Population: Study was stopped early, before outcomes could be measured, due to manufacturing issues with the study drug
Arm/Group | SCD-Omegatex™
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Days With Pain Measured by iPad Daily Report Pain Calendar
Description: as for outcome 1
Time Frame: 8 months
Population: Study was stopped early, before outcomes could be measured, due to manufacturing issues with the study drug
Arm/Group | SCD-Omegatex™
Number analyzed (Participants) | 0

5. Secondary Outcome: Changes in Individual Thermal Sensitivity Thresholds by QST
Description: as for outcome 1
Time Frame: 8 months
Population: Study was stopped early, before outcomes could be measured, due to manufacturing issues with the study drug
Arm/Group | SCD-Omegatex™
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Thrombin Generation as Assessed by Calibrated Automated Thrombogram
Description: as for outcome 1
Time Frame: 6 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: High Sensitivity C-reactive Protein (mg/L)
Description: as for outcome 1
Time Frame: 6 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Plasma Lipidomic Analysis
Description: as for outcome 1
Time Frame: 6 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Urine Resolvin D1 (pg/mg Creatinine)
Description: as for outcome 1
Time Frame: 6 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Plasma Levels of Lactate Dehydrogenase (IU/L)
Description: as for outcome 1
Time Frame: 6 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Fetal Hemoglobin (%)
Description: as for outcome 1
Time Frame: 6 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Analysis of Pro and Anti-inflammatory Cytokines in Plasma Including Interleukin (IL)1-beta, IL-4, IL-6, IL-8, IL-10 and Tumor Necrosis Factor (TNF) Alpha ( pg/ml)
Description: as for outcome 1
Time Frame: 6 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Plasma Endothelin-1(pg/ml)
Description: as for outcome 1
Time Frame: 6 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Plasma Levels Soluble Vascular Adhesion Molecule -1 (VCAM-1) (ng/ml)
Description: as for outcome 1
Time Frame: 6 months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Plasma Levels of Soluble P-selectin (ng/ml)
Description: as for outcome 1
Time Frame: 6 months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Plasma Levels of Soluble L-selectin (ng/ml)
Description: as for outcome 1
Time Frame: 6 months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Hemostatic Markers in Plasma Including D-dimers and Prothrombin Fragment 1.2 (Nmol/L)
Description: as for outcome 1
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Until one month after stopping study drug
Arm/Group | SCD-Omegatex™
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | SCD-Omegatex™ (N=3)
Mondor's disease (Reproductive system and breast disorders) | 1/1 (1) — Subject developed Mondor's disease one month after study drug was stopped due to study suspension. Admitted to hospital for one night of observation, resolved without treatment. The SAE was deemed unrelated to study medication.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | SCD-Omegatex™ (N=4)
fever (General disorders) | 1/3 (1) — influenza B, unlikely related to study medication
constipation (Gastrointestinal disorders) | 1/3 (1) — stomach cramping and constipation. Unlikely related to study medication as this was a preexisting problem.
vasoocclusive crisis (Musculoskeletal and connective tissue disorders) | 1/3 (1) — painful vasoocclusive crisis related to sickle cell disease, unlikely related to study medication
nausea (Gastrointestinal disorders) | 1/3 (1) — transient nausea, unlikely related to study medication.
stye (Eye disorders) | 1/3 (1) — stye left lower eyelid, unlikely related to study medication
rash (Skin and subcutaneous tissue disorders) | 1/3 (1) — eczematous rash, unlikely related to study drug
nosebleed (Blood and lymphatic system disorders) | 1/3 (1) — self limited, less than 5 minutes, unlikely related to study medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT02947100/Prot_SAP_000.pdf